## The Effects of Reaching Task Following Selective Trunk Stability Exercise

- NCT Number: NCT05767437
- Protocol Version:1.0
- Document Date: July 20, 2022
- Study Design: A crossover study comparing ADIM exercise and Conventional therapy
- Study Groups:
  - 1. Group A (ADIM-CT): ADIM exercise followed by Conventional therapy
  - 2. Group B (CT-ADIM): Conventional therapy followed by ADIM exercise
- Sample Size Calculation
  - Using G\*Power Version 3.1 (Franz Paul, Kiel, Germany)
  - Input parameters:
    - o Effect size: 0.44
    - $\circ$  Significance level ( $\alpha$ ): < 0.05
    - o Power: 0.80
  - Required total sample size: 12 participants

Although we initially planned to recruit 12 participants in total, considering a potential dropout rate of 10%, we recruited 10 participants per group (20 participants total)

## Statistical Analysis

- 1. Statistical Software
- Data analysis was performed using IBM SPSS 14 (version 28.0.1.1)
- 2. Tests for Normality
- The Kolmogorov-Smirnov test was used to assess data normality
- Kinematic data showed normal distribution (P > 0.05)
- 3. Basic Statistical Analysis
- Sex distribution: Chi-square test
- Comparison of demographic and clinical characteristics:

- o For normally distributed data: Independent t-test
- o For non-normally distributed data: Mann-Whitney U test (non-parametric)
- 4. Crossover Analysis
- Carryover Effect: Analysis combining data from both periods for each group
- Period Effect: Analysis of differences between groups for each treatment
- Treatment Effect: Mixed Analysis of Variance (Mixed ANOVA)
  - Factors: 2 groups × 3 assessment points
  - o Interaction analysis: Analysis of change patterns between groups over time
- 5. Multiple Comparison Adjustment
- Bonferroni correction method
- Statistical significance level: P < 0.05
- 6. Post-hoc Analysis
- Bonferroni sample t-test
- Pairwise comparisons within each group across three assessment points
- 7. Clinical Outcome Analysis
- Two-sided unpaired t-test
- Significance level: P < 0.05